CLINICAL TRIAL: NCT05973539
Title: Investigating Blood Lipid Responses to Dietary Macronutrient Content
Brief Title: Blood Lipid Responses to Diet
Acronym: BoLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 316098
Record Dates: First submitted 2023-01-09; First posted 2023-08-03 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Nutritional and Metabolic Diseases
MeSH Terms: conditions — Nutritional and Metabolic Diseases | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High carbohydrate, low fat diet (Experimental): 65% of energy is derived from carbohydrates, 20% from fat, and 15% from protein.
  Interventions: Other: Diet
- High fat, low carbohydrate diet (Experimental): 65% of energy is derived from fat, 20% from carbohydrates, and 15% from protein.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Eucaloric diet enriched in either carbohydrates or fat (both contributing to 65% total energy intake)

SUMMARY:
The macronutrient composition of our diet (proportions of carbohydrates, fats and proteins) strongly influences the way our body stores and utilises substrates (e.g., fats and sugars), which in turn influences our risk of developing cardiometabolic diseases (e.g., coronary artery disease or insulin resistance). The optimal dietary composition to lower the risk of cardiometabolic disease is unknown.

In a randomized, parallel design, this study will investigate how the overconsumption of carbohydrates and fats affects blood lipid responses and liver metabolism in adults free from metabolic disease. By genotyping participants, we will also examine the interaction between macronutrient content and an individual's genes on blood lipid responses and liver metabolism.

DETAILED DESCRIPTION:
Dietary and lifestyle interventions are central to lowering the risk and preventing the development of metabolic disease, including non-alcoholic fatty liver disease, type 2 diabetes, and cardiovascular disease. There is, however, no one fits all dietary approach, and in the context of diets where an individual is not gaining or losing weight (known as eucaloric), the optimal macronutrient composition associated with a reduced risk of metabolic disease and dyslipidemia is highly debated. For instance, eating less of one macronutrient implies eating more of another; a reduction in the intake of dietary carbohydrates is met by an increase in dietary fats. How this affects one's metabolic health in the setting when someone is not gaining or losing body weight is unclear.

Therefore, this study aims to provide an understanding of the effect that the quantity of specific dietary macronutrients (e.g., carbohydrates, fats) have on plasma triglyceride concentrations in both the fasting and postprandial state, liver fat content and metabolism, and cardiac fat content and function. We will also examine if an individual's genotype affects the metabolic response to a shift in dietary macronutrient content.

Sixty volunteers free from metabolic disease will be recruited into a randomized, parallel-armed dietary intervention study. Participants will consume either a low carbohydrate, high-fat diet or a high carbohydrate, low-fat diet for up to 28 days. Diets will be eucaloric (i.e., designed to meet the individual participant's energy requirements). Comprehensive in vivo metabolic and physiological testing will be performed before and after the experimental diet to document the effects of the overconsumption of specific macronutrients (i.e., fats or carbohydrates) on liver and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged ≥18 to ≤65 years
* Body mass index (BMI) ≥19 to ≤35 kg/m2
* No medical condition or relevant drug therapy that is known to affect the liver, adipose tissue, or cardiac metabolism.
* Weight stable for the previous 3 months

Exclusion Criteria:

* Aged <18 or >65 years
* BMI <19 or >35 kg/m2
* A blood haemoglobin <135 mg/dL for men and <120 mg/dL for women
* Donated (or lost) ≥250 mL of blood in the previous two months
* On a weight loss diet or decreased their body weight by >5% in the previous 3 months
* Currently adhering to or have consumed in the previous 3 months a diet with a notably altered macro-nutrient content (e.g. high-fat - low-carbohydrate diet)
* Have increased their body weight by >5% in the previous 3 months
* Any metabolic condition or relevant drug therapy
* Current smoker
* History of alcoholism or a greater than recommended alcohol intake (>30 g of alcohol daily for men and >20 g of alcohol daily for women)
* History of albumin allergy.
* Pregnant or nursing mothers
* History of severe claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in plasma triglyceride concentrations [mmol/L] | Pre- and post-diet [21-28 days]
  Change in plasma triglyceride concentrations in response to consumption of macronutrient meal will be measured by basic clinical chemistry before and at the end of the dietary intervention.

SECONDARY OUTCOMES:
Change in liver fat content [%] | Pre- and post-diet [21-28 days]
  Liver fat content (intra-hepatic triglyceride) will be measured before and at the end of the dietary intervention by magnetic resonance imaging/spectroscopy
Change in cardiac fat content [%] | Pre- and post-diet [21-28 days]
  Cardiac fat content will be measured before and at the end of the dietary intervention by magnetic resonance imaging/spectroscopy
Change in the contribution of dietary and adipose tissue derived fatty acids to very low density lipoprotein-triglyceride (VLDL-TG) palmitate | Pre- and post-diet [21-28 days]
  Through measuring the incorporation of [13C]palmitate and [2H2]palmitate in isolated plasma VLDL during a mixed-macronutrient feeding test.
Change in hepatic fatty acid synthesis | Pre- and post-diet [21-28 days]
  Measured by incorporation of [2H2] palmitate from 2H2O into VLDL-triglyceride
Influence of genotype on the change in plasma lipid content [mmol/L] | Pre- and post-diet [21-28 days]
  Change in plasma lipid concentrations in the fasting state and in response to consumption of macronutrient meal will be measured by basic clinical chemistry before and at the end of the dietary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Leane Hodson, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Oxford Centre for Diabetes, Endocrinology and Metabolism, University of Oxford, Oxford
  - Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD with other researchers